CLINICAL TRIAL: NCT03286751
Title: A Study to Evaluate the Pharmacokinetics and Glucodynamics of LY900014 and Humalog Across Different Subcutaneous Doses in Healthy Subjects
Brief Title: A Comparative Study of LY900014 to Insulin Lispro (Humalog) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16898; 2017-001859-32 (EudraCT Number); I8B-MC-ITSH (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY900014 (Experimental): Single dose of 7 units (U), 15 U, and 30 U of LY900014 administered subcutaneously (SC) in three of six periods.
  Interventions: Drug: LY900014
- Insulin Lispro (Humalog) (Active Comparator): Single dose of 7 U, 15 U, and 30 U of insulin lispro administered SC in three of six periods.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro — Administered SC
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro (Humalog)

SUMMARY:
This study compares LY900014, a drug that lowers blood sugar, with insulin lispro (Humalog). Both drugs are given by injection under the skin of the abdomen. The study will be conducted in healthy people to investigate how quickly and how much LY900014 is absorbed and the effect of different doses of LY900014 on blood sugar levels in comparison with insulin lispro. The study will last about 7 to 12 weeks for each participant, including screening and follow up. Screening is required within 28 days prior to entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or a female (not pregnant and agreeable to take birth control measures until one month after study completion)
* Have a body mass index (BMI) of 18 to 30 kilogram per square meter (kg/m²)
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results
* Are nonsmokers, have not smoked for at least 6 months prior to entering the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days
* Have previously participated or withdrawn from this study
* Have donated blood or have blood loss of more than 500 mL within the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Neuss

REFERENCES:
- [Derived] Leohr J, Dellva MA, Carter K, LaBell E, Linnebjerg H. Ultra Rapid Lispro (URLi) Accelerates Insulin Lispro Absorption and Insulin Action vs Humalog(R) Consistently Across Study Populations: A Pooled Analysis of Pharmacokinetic and Glucodynamic Data. Clin Pharmacokinet. 2021 Nov;60(11):1423-1434. doi: 10.1007/s40262-021-01030-0. Epub 2021 May 27. PMID 34041713
- [Derived] Leohr J, Dellva MA, LaBell E, Coutant DE, Klein O, Plum-Moerschel L, Zijlstra E, Linnebjerg H. Pharmacokinetic and Glucodynamic Responses of Ultra Rapid Lispro vs Lispro Across a Clinically Relevant Range of Subcutaneous Doses in Healthy Subjects. Clin Ther. 2020 Sep;42(9):1762-1777.e4. doi: 10.1016/j.clinthera.2020.07.005. Epub 2020 Sep 6. PMID 32900535

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 6-period crossover study in which participants received a single 7 Unit (U), 15 U, or 30 U subcutaneous (SC) dose of LY900014 or Humalog in one of six sequences. There was a washout period of ≥ 3 days between each euglycemic clamp procedure.
Groups:
- Sequence 1: ABFCED: Participants received a single SC dose in each treatment period.
  A = 7 U LY900014
  B = 15 U LY900014
  F = 30 U Humalog
  C = 30 U LY900014
  E = 15 U Humalog
  D = 7 U Humalog
- Sequence 2: BCADFE: Participants received a single SC dose in each treatment period.
  B = 15 U LY900014
  C = 30 U LY900014
  A = 7 U LY900014
  D = 7 U Humalog
  F = 30 U Humalog
  E = 15 U Humalog
- Sequence 3: CDBEAF: Participants received a single SC dose in each treatment period.
  C = 30 U LY900014
  D = 7 U Humalog
  B = 15 U LY900014
  E = 15 U Humalog
  A = 7 U LY900014
  F = 30 U Humalog
- Sequence 4: DECFBA: Participants received a single SC dose in each treatment period.
  D = 7 U Humalog
  E = 15 U Humalog
  C = 30 U LY900014
  F = 30 U Humalog
  B = 15 U LY900014
  A = 7 U LY900014
- Sequence 5: EFDACB: Participants received a single SC dose in each treatment period.
  E = 15 U Humalog
  F = 30 U Humalog
  D = 7 U Humalog
  A = 7 U LY900014
  C = 30 U LY900014
  B = 15 U LY900014
- Sequence 6: FAEBDC: Participants received a single SC dose in each treatment period.
  F = 30 U Humalog
  A = 7 U LY900014
  E = 15 U Humalog
  B = 15 U LY900014
  D = 7 U Humalog
  C = 30 U LY900014
Period: Period 1
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 7 | 7 | 7 | 7 | 7
Received at Least One Dose of Study Drug | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 7 | 7 | 7 | 6 | 7
Completed | 7 | 7 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 7 | 7 | 7 | 6 | 7
Completed | 7 | 6 | 7 | 7 | 6 | 7
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Personal Reasons | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 6 | 7 | 7 | 6 | 7
Completed | 7 | 6 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 6 | 7 | 7 | 6 | 7
Completed | 7 | 6 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 6 | 7 | 7 | 6 | 7
Completed | 7 | 6 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 4
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 6 | 7 | 7 | 6 | 7
Completed | 7 | 6 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 6 | 7 | 7 | 6 | 7
Completed | 7 | 6 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 5
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 6 | 7 | 7 | 6 | 7
Completed | 7 | 6 | 7 | 7 | 5 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 6
Arm/Group | Sequence 1: ABFCED | Sequence 2: BCADFE | Sequence 3: CDBEAF | Sequence 4: DECFBA | Sequence 5: EFDACB | Sequence 6: FAEBDC
Started | 7 | 6 | 7 | 7 | 5 | 7
Completed | 7 | 6 | 7 | 7 | 5 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Participants who received at least one dose of study drug.
Groups:
- Overall: All participants who received at least on dose of study drug.
Arm/Group | Overall
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 42

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Versus Time Curve (AUC)
Description: Pharmacokinetics: Insulin Lispro Area Under the Concentration Curve From Time Zero to 10 Hours Post Dose [AUC(0-10h)]
Time Frame: Day 1: Pre-dose, 5, 10, 15, 20, 25, 30, 35, 40, 50, 60, 70, 90, 120, 150, 180, 210, 240, 300, 360, 420, 480, 540, and 600 minutes post-dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole * hour per liter(pmol*/L)
Groups:
- 7 U Humalog: Single SC dose 7 U Humalog.
- 7 U LY900014: Single SC dose 7 U LY900014.
- 15 U Humalog: Single SC dose 15 U Humalog.
- 15 U LY900014: Single SC dose 15 U LY900014.
- 30 U Humalog: Single SC dose 30 U Humalog.
- 30 U LY900014: Single SC dose 30 U LY900014.
Arm/Group | 7 U Humalog | 7 U LY900014 | 15 U Humalog | 15 U LY900014 | 30 U Humalog | 30 U LY900014
Number analyzed (Participants) | 40 | 40 | 41 | 40 | 40 | 41
picomole * hour per liter(pmol*/L) | 649 (16) | 656 (17) | 1400 (19) | 1450 (17) | 3050 (18) | 3180 (20)
Statistical Analysis 1: Comparison: 7 U Humalog vs 7 U LY900014; Test type: Superiority; p = 0.5495, Mixed Models Analysis; Ratio of Geometric LSMeans = 1.01, 95% CI 2-sided [0.974 to 1.05]
Statistical Analysis 2: Comparison: 15 U Humalog vs 15 U LY900014; Test type: Superiority; p = 0.2236, Mixed Models Analysis; Ratio of Geometric LSMeans = 1.02, 95% CI 2-sided [0.986 to 1.06]
Statistical Analysis 3: Comparison: 30 U Humalog vs 30 U LY900014; Test type: Superiority; p = 0.0727, Mixed Models Analysis; Ratio of Geometric LSMeans = 1.03, 95% CI 2-sided [0.997 to 1.07]

2. Secondary Outcome: Glucodynamics: Total Amount of Glucose Infused (Gtot)
Description: Glucodynamics: Total Amount of Glucose Infused (Gtot) Over the Duration of Clamp
Time Frame: Day 1: Every minute starting from the pre-dose and throughout the duration of the clamp until 10 hours post-dose
Population: All participants who received at least one dose of study drug and completed at least one clamp procedure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per kilogram (mg/kg)
Arm/Group | 7 U Humalog | 7 U LY900014 | 15 U Humalog | 15 U LY900014 | 30 U Humalog | 30 U LY900014
Number analyzed (Participants) | 40 | 40 | 41 | 40 | 40 | 41
milligrams per kilogram (mg/kg) | 1120 (53) | 1080 (60) | 1970 (44) | 1860 (45) | 3290 (32) | 3030 (36)
Statistical Analysis 1: Comparison: 7 U Humalog vs 7 U LY900014; Test type: Superiority; p = 0.5749, Mixed Models Analysis; Ratio of Geometric LSMeans = 0.97, 95% CI 2-sided [0.87 to 1.08]
Statistical Analysis 2: Comparison: 15 U Humalog vs 15 U LY900014; Test type: Superiority; p = 0.1578, Mixed Models Analysis; Ratio of Geometric LSMeans = 0.92, 95% CI 2-sided [0.83 to 1.03]
Statistical Analysis 3: Comparison: 30 U Humalog vs 30 U LY900014; Test type: Superiority; p = 0.1351, Mixed Models Analysis; Ratio of Geometric LSMeans = 0.92, 95% CI 2-sided [0.83 to 1.03]

ADVERSE EVENTS:
Time Frame: Baseline to study completion (up to 12 weeks)
Groups:
- 30 U Humalog: Single SC dose 15 U Humalog.
Arm/Group | 7 U LY900014 | 15 U LY900014 | 30 U LY900014 | 7 U Humalog | 15 U Humalog | 30 U Humalog
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/41 | 0/40 | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/41 | 0/40 | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 7/40 | 5/40 | 14/41 | 8/40 | 6/41 | 5/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7 U LY900014 (N=40) | 15 U LY900014 (N=40) | 30 U LY900014 (N=41) | 7 U Humalog (N=40) | 15 U Humalog (N=41) | 30 U Humalog (N=40)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 6 (6) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 4 (4) | 6 (6) | 8 (8) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03286751/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT03286751/SAP_001.pdf